CLINICAL TRIAL: NCT06188598
Title: Time-restricted Eating as a Dietary Intervention for Dyslipidemia in Peri- and Postmenopausal Women
Brief Title: Time-restricted Eating in Peri- and Postmenopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Leilah Kristine Grant, Investigator, Instructor in Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022P002288
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Dyslipidemias; Obesity; Menopause
MeSH Terms: conditions — Dyslipidemias; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized on 1:1 bases to time-restricted eating or unrestricted eating
Who Masked: Outcomes Assessor
Masking Description: Blood tests and assays, DXA scans, body weight, vitals, etc. are performed by assessors blinded to the condition and aims of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted eating (TRE) (Experimental): Participants in the TRE group are instructed to restrict eating to an 8-hr window but were not asked to change the type or amount of food typically consumed. The 8-hour window (e.g., 10am - 6pm) has to be the same each day starting at least 2 hours after wake and ending at least 2 hours before bed.
  Interventions: Behavioral: Time-restricted eating
- Unrestricted eating (No Intervention): Participants are instructed to continue their diet as normal without changing the type, amount or timing of food typically consumed.

INTERVENTIONS:
Behavioral: Time-restricted eating — Eating is restricted to an 8-hour window that is the same each day (e.g., 10am - 6pm)
  Arms: Time-restricted eating (TRE)

SUMMARY:
The overall objective of the study is to examine the effect of an 8-hour time-restricted eating intervention on lipid levels and body composition in peri- and recently postmenopausal women with untreated dyslipidemia.

DETAILED DESCRIPTION:
This is a randomized controlled trial investigating the effects of an 8-TRE intervention compared to ad libitum eating (control) on metabolic health and body composition in recently postmenopausal women with untreated dyslipidemia. Following a 1-week baseline assessment, participants will be randomized to either a TRE or unrestricted control diet schedule (1-to-1 ratio) for 8 weeks. At baseline and weeks 4 and 8 of the intervention, daily eating and sleep patterns will be assessed for one week, followed by collection of fasting lipids and metabolic labs, body weight and vital signs; questionnaires assessing sleep and mood health, actigraphy and body composition via whole-body dual-energy x-ray absorptiometry will be assessed at baseline and week 8.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 40-58 years
* Perimenopausal or recently postmenopausal, >1 year and <5 years
* BMI > 30 kg/m2
* Dyslipidemic, defined as the presence of one or more lipid-based cardiovascular disease risk-enhancing factors per American College of Cardiology/American Heart Association guidelines
* Normal renal and hepatic function
* Perimenopausal women, a negative pregnancy test

Exclusion Criteria:

Dietary factors:

* Diagnosis, or strong clinical suspicion, of eating disorders, including but not limited to, anorexia nervosa, bulimia nervosa, binge eating disorder
* Concurrent dietary intervention or modification unrelated to study procedures

Psychiatric factors:

* Current major depressive episode
* Suicidal ideation
* Lifetime history of bipolar disorder, psychosis, or other serious mental health problem
* Current alcohol/substance use disorder

Medical factors:

* Use of lipid-lowering or lipid-enhancing medications
* Use of systemic hormonal (estrogens and/or progestin) therapies
* Use of weight loss medications or supplements
* Use of medications that may cause weight loss or gain, unless body weight and medication usage remained stable for at least 6 months
* Previous weight loss surgery
* Abnormal vital signs at screening visit
* Body weight > 350 pounds, per DXA scan limits
* Malignancy within past 2 years
* Major surgery within past 3 months
* Medical instability considered to interfere with study procedures
* Contraindications to DXA scanning
* Use of medications that have the potential to cause hypoglycemia (e.g., insulin, sulfonylureas)
* Undergoing treatment for cancer
* Use of medications for which time-restricted eating would interfere with recommended timing of medication ingestion with food intake.

Lifestyle and other factors:

* Irregular sleep/wake schedule
* Shiftwork
* Recent travel across 2 or more time zones
* Recent change in exercise habits
* Work or social schedules that would impede ability to adhere to study protocol

Adherence factors:

-Inability to adhere to study procedures completed between screening and randomization visits

Off-Study Criteria:

* Initiation of new medications for lipid management, weight loss, hormonal medications, or other medications that may cause changes in weight or lipid levels
* Development of any significant medical problem
* Enrollment in another clinical trial involving study procedures or medications that might interfere with study procedures.
* Significant deviation from study protocol or protocol violation
* Inability to adhere to time-restricted eating window

Ages: 40 Years to 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2024-12-21 (Estimated); Study Completion 2024-12-21 (Estimated)

PRIMARY OUTCOMES:
Change in fasting triglyceride levels | Baseline (week 0) and post-intervention (week 8)
  Pre- to post-intervention change in fasting triglyceride levels (mg/dL)
Change in visceral adiposity | Baseline (week 0) and post-intervention (week 8)
  Pre- to post-intervention change in visceral adiposity (mass) as measured by dual energy x-ray absorptiometry scan

SECONDARY OUTCOMES:
Change in body weight | Baseline (week 0) and post-intervention (week 8)
  Pre- to post-intervention change in body weight (kg)
Change in high-density lipoprotein cholesterol (HDL-C) | Baseline (week 0) and post-intervention (week 8)
  Pre- to post-intervention change in HDL-C (mg/dL)
Change in low-density lipoprotein cholesterol (LDL-C) | Baseline (week 0) and post-intervention (week 8)
  Pre- to post-intervention change in LDL-C (mg/dL)
Change in systolic blood pressure | Baseline (week 0) and post-intervention (week 8)
  Pre- to post-intervention change in systolic blood pressure (mmHg)
Change in sleep quality | Baseline (week 0) and post-intervention (week 8)
  Change in sleep quality as measure by the Pittsburgh Sleep Quality Index (PSQI) global score. PSQI global score range is 0-21 with higher scores indicating more sleep disturbance.
Change in depressive symptoms | Baseline (week 0) and post-intervention (week 8)
  Change in depressive symptoms as measure by the Patient Health Questionnaire-8 (PHQ-8). The PHQ-8 score ranges from 0-24 with higher scores indicating greater depressive symptoms.
Change in positive and negative affect | Baseline (week 0) and post-intervention (week 8)
  Change in positive and negative affect as measure by the Positive and Negative Affect Schedule. The PANAS Positive and Negative scores range from 10-50 with higher scores indicating greater postive and negative affect, respectively.
Change in sleep duration | Assessed daily over 1 week at baseline (week 0) and post-intervention (week 8)
  Change in sleep duration based on the average of self-reported sleep duration over 1 week
Change in sleep efficiency | Assessed daily over 1 week at baseline (week 0) and post-intervention (week 8)
  Change in sleep efficiency based on the average of self-reported sleep efficiency over 1 week. Sleep efficiency to be calculated as total sleep time/ time in bed.

OTHER OUTCOMES:
Time-course of triglyceride levels across 8 weeks | Baseline (week 0), mid- (week 4) and post-intervention (week 8)
  The time course of triglyceride (mg/dL) levels measured pre- mid- and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Leilah K Grant, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No